CLINICAL TRIAL: NCT00333918
Title: Efficacy and Safety Study of Topical Bromfenac Ophthalmic Solution vs. Placebo for Treatment of Ocular Inflammation and Pain Associated With Cataract Surgery
Brief Title: Safety/Efficacy of Bromfenac Ophthalmic Solution for Ocular Inflammation and Pain Associated With Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISTA-BR-CS02
Record Dates: First submitted 2006-06-04; First posted 2006-06-06 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Pain; Inflammation
Keywords: Cataract Extraction; Anti-Inflammatory Agents, Non-Steroidal
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1-bromfenac ophthalmic solution (Experimental): sterile ophthalmic solution
  Interventions: Drug: bromfenac ophthalmic solution
- 2-placebo comparator (Placebo Comparator): sterile ophthalmic solution
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: bromfenac ophthalmic solution
  Arms: 1-bromfenac ophthalmic solution
Drug: placebo comparator
  Arms: 2-placebo comparator

SUMMARY:
The primary objective of this study is to investigate the efficacy and safety of bromfenac ophthalmic solution for treatment of ocular inflammation and pain in subjects who undergo cataract extraction and intraocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral cataract surgery with no other ophthalmic surgical procedures planned during cataract surgery
* Agree to return for all required visits
* Agree to avoid disallowed medications

Exclusion Criteria:

* Known hypersensitivity to bromfenac and salicylates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2006-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Reduction of ocular inflammation

SECONDARY OUTCOMES:
Secondary efficacy outcome for ocular pain will be the proportion of treated subjects that are pain free

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Bianca, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- Irvine, California, United States